CLINICAL TRIAL: NCT03618082
Title: Effect of Targeted Analgesia to ANI (Analgesia/ Nociception Index) During General Anesthesia on Immediate Postoperative Pain and Perioperative Hemodynamic: Multicenter Randomized Controlled Study
Brief Title: GOAL-Directed ANalgesia (GOALDAN)
Acronym: GOALDAN
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Fondation Apicil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CHU-401; 2017-A03268-45 (Other: 2017-A03268-45)
Record Dates: First submitted 2018-07-18; First posted 2018-08-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Immediate Severe Postoperative Pain; Perioperative Hemodynamic
Keywords: prospective; single blind; multicenter; randomized; controlled; Analgesia Nociception Index (ANI); Postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Randomization in 2 groups 1- control group : patients receiving a general anesthesia with propofol, ketamine and remifentanil with or without curare for the induction, desflurane, remifentanil (curare or not) for the maintenance, the dosage of the anesthetic agents will be decided by the anesthesiologist responsible for the patient based on the usual practice. 2- experimental group : patients receiving a general anesthesia with propofol, ketamine and remifentanil with or without curare for the induction, desflurane, remifentanil (curare or not) for the maintenance, administered according to a specific algorithm. In this group, the remifentanil administration will be piloted by the ANI (50 to 80), as well as the prophylactic administration of morphine at the end of the intervention. Administration of 2mg of morphine immediately before the extubating if ANI<50. And, desflurane will be administered with a targeted purpose of 0.8 to 1.2 MAC.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- usual practice (Active Comparator): control group (usual practice): patients receiving a general anesthesia with propofol, ketamine and remifentanil with or without curare for the induction, and desflurane and remifentanil (with or without curare) for the maintenance. The dosage of the anesthetic agent, as well as the prophylactic administration of morphine at the end of the intervention, will be decided by the anesthesiologist.
  Interventions: Drug: Anesthesic agent guided by ANI (Interventional Group); Drug: Administration of the lowest effective concentration of desflurane (Interventional Group)
- targeted analgesia to ANI (Experimental): experimental group: patients receiving a general anesthesia with propofol, ketamine and remifentanil with or without curare for the induction, and desflurane and remifentanil (with or without curare) for the maintenance, as well as the prophylactic administration of morphine at the end of the intervention, will be administered according to the ANI.
  - In addition, desflurane will be administered with a targeted purpose of minimal alveolar concentration (MAC).
  Interventions: Drug: Anesthesic agent guided by ANI (Interventional Group); Drug: Administration of the lowest effective concentration of desflurane (Interventional Group)

INTERVENTIONS:
Drug: Anesthesic agent guided by ANI (Interventional Group) — Anesthesic agent guided by ANI (Interventional Group) The remifentanil administration will be piloted by the ANI, as well as the prophylactic administration of morphine at the end of the intervention.
Drug: Administration of the lowest effective concentration of desflurane (Interventional Group) — Administration of the lowest effective concentration of desflurane (Interventional Group) Desflurane will be administered with a targeted purpose of minimal alveolar concentration (MAC).

SUMMARY:
The primary purpose of GOALDAN study is to demonstrate the superiority of a targeted perioperative analgesic strategy by the ANI over the usual practice on the incidence of immediate postoperative pain.

The investigators hypothesized that a prophylactic administration of morphine in patients with risk of postoperative pain determined by the ANI at the end of the intervention would reduce the incidence of immediate postoperative pain and that the targeted analgesia to ANI and minimal alveolar concentration (MAC) of desflurane could improve the perioperative hemodynamic, and the postoperative becoming.

DETAILED DESCRIPTION:
Visits:

* The patient will arrive in the department the day before the surgical intervention (D-1). During this preoperative visit (D-1), the investigator

  * will preselect potentially eligible patients
  * will offer to participate to this study
  * will give the notice form to the patients
  * will present the research: objectives, benefits and constraints for the patients
  * will check that patients understand the verbally administered Numeric Rating Scale (NRS) for the assessment of the postoperative This verbally administered NRS is routinely presented to all patients at a surgical intervention.
* The intervention day (D0):

The investigator will collect the signed consent form after having ascertained the understanding of the notice form by the patient and checking the inclusion and non-inclusion criteria.

The randomization will be done via the eCRF module (allocation group and number) and the preoperative data registration in the eCRF.

• Surgical intervention (D0): All patients will receive a usual multimodal analgesia associating level 1 analgesics (acetaminophen, ketoprofen, nefopam) or level 2 (tramadol) administered 30 to 60 min before the foreseeable end of the surgical intervention. All patients will receive 0.1 to 0.2 mg/kg of morphine within the 30 min preceding the end of the surgical intervention according to the usual practice.

Once the patient transferred to the recovery room, the assessment of the primary outcome (verbally administered NRS) will be done by the nurse responsible for the patient, when the patient arrives, during the stay and when the patient leaves the recovery room. If the verbally NRS > 3, a morphine titration by IV administration of 2 to 3 mg of morphine will be realised then the verbally NRS will be collected 5 min after, according to the usual practice. This morphine titration will continued until the obtaining of a verbal NRS ≤ 3.

As an alternative to this morphine titration, where possible, a peripheral nerve block may be proposed to the patient and performed by the investigator to relieve the patient.

If the patient is transferred directly in ICU without being extubated at the end of the intervention and so without transiting by the recovery room, the patient will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* 18≤ Age <65 years old
* Patient operated on a scheduled surgery under general anesthesia
* Patient with a American Society of Anesthesiologists (ASA) score of I to III
* Patient having given his consent in the manner described in Article L1122-1-1 of the Public Health Code
* Patient affiliated with a social security regimen or beneficiary of such a regimen

Exclusion Criteria:

* general anesthesia without extubating (laryngeal mask)
* neuraxial preoperative regional anesthesia (epidural or rachianalgesia)
* opioid-free anesthesia
* preoperative peripheral nerve block with analgesic aim (infiltration of a local surgical anesthetic or transversus abdominis plane block-TAP block-authorized)
* arrhythmia or the presence of a pacemaker
* ambulatory surgery
* cardiac or cerebral surgery
* obstetrical surgery (caesarean)
* surgery performed with neuraxial regional anesthesia or peripheral anesthesia alone
* surgery performed in prone position
* urgent surgery
* endoscopic procedure or interventional radiology
* chronic pain treated with opiates
* expected surgery duration < 1h
* pathology of the autonomic nervous system (epilepsy, history of transient attack or stroke, paraplegia, hemiplegia, orthostatic hypotension, autonomic dysfunction)
* Patient with cardiogenic or septic shock
* Continuous infusion of vasoactive agents (ephedrine, phenylephrine, adrenaline, or noradrenaline)
* Postoperative transfer planned in intensive care unit (intubated patient) after surgery
* Person under tutorship or curatorship
* Pregnancy
* Breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2019-06-06 (Actual); Primary Completion 2022-05-13 (Estimated); Study Completion 2022-08-13 (Estimated)

PRIMARY OUTCOMES:
immediate maximum postoperative pain in recovery room defined by a score > 3 on a verbally administered numeric rating scale (NRS) variating from 0 to 10. | From day 0 to day 28
  Once the patient transferred to the recovery room, the assessment of the primary outcome (verbally administered NRS) will be done by the nurse responsible for the patient, when the patient arrives, during the stay and when the patient leaves the recovery room

SECONDARY OUTCOMES:
Maximum pain score during the first postoperative day (numeric rating scale variating from 0 to 10). | every 6 hours during the 24 first hours.
  The patient chooses on a scale numeric range a number between 0 and 10 to characterise the intensity of the pain during the first postoperative day : 0 if the pain is mild (better outcome), 10 if the pain is severe (worse outcome).This numeric rating scale will be assessed every 6 hours during the 24 first hours (H0 = arrival hour at the recovery room).
Score Postoperative D1 Pain Management (numeric rating scale variating from 0 to 10) | At day 1
  The patient chooses on a scale numeric range from 0 to 10, a number which characterises the overall satisfaction of pain management : if the pain management is correct (10) or if the pain management is not correct (0).
dose of morphine in the recovery room | At day 0
  will be compared between groups by test t of Student or test not parametrize of Mann-Whitney if the conditions of the test t are not respected (study of the normality, homoscedasticity studied by test of Fisher-Snedecor). The results will be expressed in terms of size of effect and reliable interval in associated 95 %. These analyses can be secondly completed, in multivariate situation, by models of regression of linear type; covariables will be considered with regard to the clinical relevance and the results of analyses univariate preliminary. The results will be expressed in terms of coefficients of regression and reliable intervals in associated 95 %.
postoperative nausea and vomiting in the recovery room | At day 1
  In both groups, the prevention of the nausea and the vomitings will be administered according to the current recommendations (dexamethasone 4 mg and droperidol 0,625-1,25 mg it peroperatoire at the patients at risk, defined by a score of Apfel 2). In case of NVPO during the first 24 post-operative hours, the administration of 4 mg of ondansétron will be realized, according to the recommendations.
total dose of morphine during the first postoperative day (mg) | At day 1
  will be compared between groups by test t of Student or test not parametrique of Mann-Whitney if the conditions of the test t are not respected (study of the normality, homoscedasticity studied by test of Fisher-Snedecor). The results will be expressed in terms of size of effect and reliable interval in associated 95 %. These analyses can be secondly completed, in multivariate situation, by models of regression of linear type; covariables will be considered with regard to the clinical relevance and the results of analyses univariées preliminary. The results will be expressed in terms of coefficients of regression and reliable intervals in associated 95 %.
regional anesthesia for postoperative analgesic purposes | At day 1
the duration in the recovery room (time to obtain an Aldrete score ≥9) (min) | From day 0 to day 28
  will be compared between groups by test t of Student or test not parametrize of Mann-Whitney if the conditions of the test t are not respected (study of the normality, homoscedasticity studied by test of Fisher-Snedecor). The results will be expressed in terms of size of effect and reliable interval in associated 95 %. These analyses can be secondly completed, in multivariate situation, by models of regression of linear type; covariables will be considered with regard to the clinical relevance and the results of analyses univariées preliminary. The results will be expressed in terms of coefficients of regression and reliable intervals in associated 95 %.
destination of the patient after surgery (unit of surgery, continuous care, resuscitation). | From day 0 to day 28
  Test of chi² or exact test of Fisher if necessary. Secondly, this analysis can be completed, in multivariate situation, by a mixed generalized linear model of logistic type allowing to take into account variability inter and intracentre. Covariables will be considered with regard to the clinical relevance (other treatments, use of vasopresseurs continuous, type of surgery) and results of analyses univariate preliminary. The results will be expressed in terms of reports of the quotations and the reliable intervals in associated 95 %.
incidence of postoperative complications on the first and seventh postoperative days for hospitalized patients using Post-Operative Morbidity Survey (POMS). | From day 0 to day 1 and until day 7
  Post-operative complications in the first and seventh day post-operative will be compared by test of chi² or where necessary, by the exact test of Fisher.
  Secondly, this analysis can be completed, in multivariate situation, by a mixed generalized linear model of logistic type allowing to take into account variability inter and intracentre. Covariables will be considered with regard to the clinical relevance (other treatments, use of vasopresseurs continuous, type of surgery) and results of analyses univariées preliminary. The results will be expressed in terms of reports of the quotations and the reliable intervals in associated 95 %.
duration of the hospitalization (day) | From day 0 to day 28
  Duration of hospitalization will be compared between groups by test t of Student or test not paramétrique of Mann-Whitney if the conditions of the test t are not respected (study of the normality, homoscédasticité studied by test of Fisher-Snedecor). The results will be expressed in terms of size of effect and reliable interval in associated 95 %. These analyses can be secondly completed, in multivariate situation, by models of regression of linear type; covariables will be considered with regard to the clinical relevance and the results of analyses univariées preliminary. The results will be expressed in terms of coefficients of regression and reliable intervals in associated 95 %.
Mortality at Day 28 | At day 28
  The survival to day 28 comment surgery will be estimated(esteemed) by curve of Kaplan-Meier and compared between groups of randomization by test of the log-rank in univariate situation and model of Cox in multivariated analysis. The results will be expressed in terms of relationship of immediate risks and reliable intervals in associated 95 %.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Etienne BAZIN, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, Auvergne, France

REFERENCES:
- [Derived] Michalot A, Bazin JE, Richebe P, Allaouchiche B, Boselli E. Effect of GOAL-Directed ANalgesia using ANI (Analgesia/Nociception Index) during general anesthesia on immediate postoperative pain and intraoperative hemodynamics in adult patients (GOALDAN study): a study protocol for randomized, controlled, multicenter trial. Trials. 2022 Apr 25;23(1):353. doi: 10.1186/s13063-022-06273-1. PMID 35468803